CLINICAL TRIAL: NCT06142643
Title: Safety and Effectiveness Clinical Evaluation of Range of Injectable Medical Devices Viscol in Aesthetic Treatment
Brief Title: Safety and Effectiveness Clinical Evaluation of Injectable Medical Devices Viscol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kylane Laboratoires (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23E1077
Record Dates: First submitted 2023-11-02; First posted 2023-11-21 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Aesthetic Dermatology
Keywords: Aesthetic; dermatology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device under investigation (Experimental)
  Interventions: Device: Dermal Filler Device

INTERVENTIONS:
Device: Dermal Filler Device — Injection of the device by investigators according to the IFU

SUMMARY:
Evaluation of safety and performance of HA based injectable device for skin quality improvement

DETAILED DESCRIPTION:
The primary objective is to evaluate the effectiveness of the device used one month (M1) after treatment using clinical evaluation of the global aesthetic improvement (GAIS) rated by an independent investigator.

The secondary objectives of the study are to collect data on:

* the effectiveness four months (M4) after treatment.
* the effectiveness on the improvement of facial skin quality by objective measurements of skin biomechanical parameters using Cutometer® and skin hydration using Moisturemeter®.
* subject's satisfaction and subject's opinion on aesthetic improvement.
* the injector's satisfaction on the injection quality.
* the safety using clinical evaluation of the Injection Site Reactions (ISR).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Subject.
2. Sex: male or female.
3. Age: between 35 and 70 years.
4. Subject seeking an improvement for HA skin quality improvement product.
5. Subject with BMI <30.
6. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study.
7. Subject having given his/her free, express, and informed consent.
8. Subject psychologically able to understand the information related to the study, and to give their written informed consent.
9. Subject registered with a social security scheme.
10. Women of childbearing potential should use a contraceptive method considered effective since at least 12 weeks and throughout the study

Exclusion Criteria:

In terms of population

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
3. Subject in a social or sanitary establishment.
4. Subject suspected to be non-compliant according to the investigator's judgment.
5. Subject having received a total of 6.000 euros as compensations for their participation in clinical research in the last 12 months, including their participation in the present study.
6. Subject enrolled in another study or whose non-enrollment period is not over.
7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up…). In terms of associated pathology
8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.
9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria …) in the 6 months before screening visit.
11. Subject with a history of streptococcal disease or an active streptococcus infection.
12. Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kylane Laboratoires, Plan-les-Ouates, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Indication
Groups:
- Viscol Face: Dermal Filler Device: Injection of the device by investigators according to the IFU in Face area
- Viscol Body: Dermal Filler Device: Injection of the device by investigators according to the IFU in Body area
Period: Overall Study
Arm/Group | Viscol Face | Viscol Body
Started | 64; 64 Indication | 22; 31 Indication
Completed | 64; 64 Indication | 22; 31 Indication
Not Completed | 0; 0 Indication | 0; 0 Indication

BASELINE CHARACTERISTICS:
Groups:
- Viscol Face: Injection of the device by investigators according to the IFU in the Face area
- Viscol Body: Injection of the device by investigators according to the IFU in the Body area
- Total: Total of all reporting groups
Arm/Group | Viscol Face | Viscol Body | Total
Number analyzed (Participants) | 64 | 22 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 22 | 86
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 53 [35 to 70] | 57 [36 to 70] | 54 [35 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 21 | 76
  Male | 9 | 1 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 64 | 22 | 86

OUTCOME MEASURES:

1. Primary Outcome: Performance at 1 Month Investigator Overall VISCOL Range
Description: Primary endpoint was the percentage of subjects having an improvement of the zone treated with the overall FILLGEL range of devices, in all the indications, as assessed by the independent investigator, one month after treatment, using the GAIS (subjects with a GAIS "improved", "much improved" or "very much improved"). This proportion of responders was compared to a theoretical proportion of 60%.
Time Frame: 1 month
Population: Primary endpoint was the percentage of subjects having an improvement of the zone treated with the overall FILLGEL range of devices, in all the indications
Measure: Count of Participants; unit: Participants
Groups:
- Viscol Face and Body: All study participants
Arm/Group | Viscol Face and Body
Number analyzed (Participants) | 86
Participants | 77
Statistical Analysis 1: Comparison: Viscol Face and Body; Test type: Other — A responder was defined by subjects with a score 1 (very much improved), 2 (much improved) or 3 (improved) on the GAIS. Inferential analysis for the primary evaluation criterion For the derived outcome responder rate at M1 (1 month after injection) for the GAIS Investigator, a binomial exact test (bilateral approach) vs 60% was applied for the overall score. This test compared the proportion of improvement to 60%; p < 0.0001, t-test, 2 sided — Power of 80%, significant result (alpha = 5%); Null hypothesis stated that less than 60% of subjects were responders with GAIS. Under the alternative hypothesis, 75% of subjects were responders

2. Secondary Outcome: Performance at 4 Months Investigator Overall VISCOL Range
Description: Percentage of responders (subjects with a GAIS "improved", "much improved" and "very much improved") for the whole VISCOL range.
Time Frame: 4 months
Population: 1 subject missed the 4 month visit. But come back for the end of the study. This is included in deviations, and has been assessed as minor deviation.
Measure: Count of Participants; unit: Participants
Arm/Group | Viscol Face and Body
Number analyzed (Participants) | 85
Participants | 69
Statistical Analysis 1: Comparison: Viscol Face and Body; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, t-test, 2 sided — Power of 80%, significant result (alpha = 5%); [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Indications With Response: GAIS Investigator Overall VISCOL Range
Description: Responder rate for the whole indication of VISCOL range at M1 and M4- GAIS investigator (N=95 indications).
  Percentage of responders (subjects with a GAIS "Very Much Improved", "Much Improved" or "Improved") for the whole VISCOL range as assessed by an independent investigator.
Time Frame: 1 month & 4 months
Population: 1 subject missed the 4 month visit. But come back for the end of the study. This is included in deviations, and has been assessed as minor deviation. Responder rate for the whole indication (N=95 indications) of VISCOL range at M1 and M4.
Measure: Number; unit: percentage of indications
Units Other Than Participants: Indications
Arm/Group | Viscol Face and Body
Number analyzed (Participants) | 64
Number analyzed (Indications) | 95
percentage of indications
  At 1 month | 85
  At 4 months | 78

4. Secondary Outcome: Performance at 1 & 4 Months Subject Overall VISCOL Range
Description: Percentage of responders for the whole VISCOL range as assessed by the subject. This percentage of responders was compared to a theoretical proportion of 60%
Time Frame: 1 month, 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Viscol Face and Body
Number analyzed (Participants) | 86
Participants
  1 month | 69
  4 months | 62

5. Secondary Outcome: Percentage of Indications With Response: GAIS Subject Overall VISCOL Range
Description: Responder rate for the whole indication of VISCOL range at M1 and M4- GAIS subject (N=95 indications) Percentage of responders (subjects with a GAIS "Very Much Improved", "Much Improved" or "Improved") for the whole VISCOL range as assessed by the subject.
Time Frame: 1 month & 4 months
Population: as for outcome 3
Measure: Number; unit: percentage of indications
Units Other Than Participants: Indication
Groups:
- Device Under Investigation 1 Month: Dermal Filler Device: Injection of the device by investigators according to the IFU at 1 month
Arm/Group | Device Under Investigation 1 Month
Number analyzed (Participants) | 64
Number analyzed (Indication) | 95
percentage of indications
  At 1 month | 80
  At 4 months | 70

6. Secondary Outcome: Percentage of Responder With Response: GAIS Investigator by Indication Overall VISCOL Range
Description: Responder rate for the whole VISCOL range by indication at M1 and M4- GAIS combined score (investigator and subjects) (N=95 indications).
  It represents the percentage of responders (subjects with a GAIS "Very Much Improved", "Much Improved" or "Improved") for the whole VISCOL range by indication as assessed by the subject as well as by the investigator.
Time Frame: 1 month & 4 months
Population: Responder rate for the whole VISCOL range by indication (N=95 indications) at M1 and M4- GAIS combined score (investigator and subjects).
  1 subject missed the 4 month visit. But come back for the end of the study. This is included in deviations, and has been assessed as minor deviation.
Measure: Number; unit: percentage of responders
Units Other Than Participants: Indications
Arm/Group | Viscol Face and Body
Number analyzed (Participants) | 86
Number analyzed (Indications) | 95
percentage of responders
  At 1 month | 73
  At 4 months | 64

7. Secondary Outcome: Injector Satisfaction Questionnaire Viscol
Description: Distribution of each item of the questionnaire answered by the injectors. For each item of the injector questionnaire, the percentage of answers "very satisfied" and satisfied were computed as "Satisfied" and the percentage of answers "Neither satisfied" ,or "dissatisfied", "dissatisfied" and "very dissatisfied" were computed as Dissatisfied.
  The measure reported is the percentage of participants who were "Satisfied".
Time Frame: D0 (Immediatly after injection)
Measure: Number; unit: percentage of participants
Arm/Group | Viscol Face | Viscol Body
Number analyzed (Participants) | 64 | 22
percentage of participants
  Ease of removal of the tip-cap | 100 | 100
  Ease of needle/cannula assembly with the syringe | 100 | 100
  Ease of injection (including extrusion force control) | 100 | 51.7
  Handling comfort | 100 | 100
  Ease of product positioning | 100 | 100
  Immediate result | 100 | 96.5
  Result after massage | 96.9 | 100

8. Secondary Outcome: Subject Satisfaction Questionnaire Viscol
Description: Distribution of each item of the questionnaire answered by the subjects injected with Viscol. For each item of the subject questionnaire, the percentage of answers "totally agree" and "agree" were computed as "Agree" and the percentage of answers "Neither agree and disagree",or "disagree" and "totally disagree" and "very dissatisfied" were computed as "Disagree".
  The measure reported is the percentage of participants who "Agree".
Time Frame: 1 month, 4 months
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Viscol Face | Viscol Body
Number analyzed (Participants) | 64 | 22
percentage of subjects
  Improvement in skin firmness at 1 month | 64.1 | 63.6
  Improvement of skin elasticity/pliability at 1 month | 76.2 | 68.2
  Improvement in skin laxity at 1 month | 51.6 | 59.1
  Improvement in skin hydration at 1 month | 70.3 | 63.6
  Improvement in skin roughness at 1 month | 53.1 | 47.6
  Improvement in skin smoothness at 1 month | 68.8 | 63.6
  Contour remodelled and more defined at 1 month | 54.7 | 31.8
  Lifting effect at 1 month | 57.1 | 50
  Improvement of skin radiance at 1 month | 68.8 | NA — This question has not been asked to subject for Viscol Body, it is not relevant
  Decrease of skin fine lines at 1 month | 65.6 | 59.1
  Improvement of the aspect of skin pores at 1 month | 67.2 | 50
  I am satisfied with the result obtained at 1 month | 79.7 | 68.2
  Improvement in skin firmness at 4 months | 68.3 | 68.2
  Improvement of skin elasticity/pliability at 4 months | 68.3 | 68.2
  Improvement in skin laxity at 4 months | 49.2 | 54.5
  Improvement in skin hydration at 4 months | 73 | 68.2
  Improvement in skin roughness at 4 months | 65.1 | 54.5
  Improvement in skin smoothness at 4 months | 74.6 | 57.1
  Contour remodelled and more defined Contour remodelled and more defined at 4 months | 47.6 | 27.3
  Lifting effect at 4 months | 54 | 50
  Improvement of skin radiance at 4 months | 69.8 | NA — This question has not been asked to subject for Viscol Body, it is not relevant
  Decrease of skin fine lines at 4 months | 61.9 | 40.9
  Improvement of the aspect of skin pores at 4 months | 69.8 | 36.4
  I am satisfied with the result obtained I am satisfied with the result obtained at 4 months | 68.3 | 38.2

9. Secondary Outcome: Percentage of Participants Experiencing Adverse Events
Description: Percentage of participants who experienced at least one Adverse Event (AE), Adverse Device Effect (ADE), and/or Serious Adverse Event (SAE)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Viscol Face | Viscol Body
Number analyzed (Participants) | 64 | 22
Participants
  At least one AE | 26 | 6
  At least one ADE | 4 | 0
  At least one SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Viscol Face | Viscol Body
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/22
Other Adverse Events (participants affected / at risk) | 26/64 | 6/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viscol Face (N=64) | Viscol Body (N=22)
Side effect (Surgical and medical procedures) | 26 (55) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT06142643/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT06142643/ICF_001.pdf